CLINICAL TRIAL: NCT01119547
Title: The Effect of Including Exercise in an Education Program for Patients With Osteoarthritis in Primary Health Care
Brief Title: Patient Education Program for Osteoarthritis With Exercise Included
Acronym: PEPOA-E
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator no longer at LU.
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEPOA-E
Record Dates: First submitted 2010-04-29; First posted 2010-05-07 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2010-04

CONDITIONS: Osteoarthritis
Keywords: Musculoskeletal Diseases; Osteoarthritis; Joint Diseases; Arthritis; Rheumatic Diseases
MeSH Terms: conditions — Osteoarthritis; Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home exercise (Experimental): The patients is training at home during 6 v. with an individual exercise program.
  Interventions: Other: Home exercise
- Exercise in group (Experimental): The patients is doing their individual exercise program in a group.
  Interventions: Other: Exercise in a group

INTERVENTIONS:
Other: Exercise in a group — The patient do their individual exercise program in a group.
  Arms: Exercise in group
Other: Home exercise — The patient exercise their individual program at home during 6 v.
  Arms: Home exercise

SUMMARY:
The purpose of this study is to investigate if inclusion of exercise in an education program for patients with osteoarthritis can improve self efficacy, self-perceived health and function.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative disease, considered to be one of the major national diseases that cause suffering for affected patients and costs for society.The predominant symptoms are pain, stiffness and impaired quality of life, often together with psychological distress. Treatment often consists of medication. Later in the disease, when the joint is destroyed, joint replacement surgery commonly occurs. Physical exercises aimed to increase muscle strength, endurance, proprioception and stability have proved to influence cartilage as well as function, symptoms and quality of life positively. Physical exercise may also reduce the need for hospital care after knee joint replacement.Research suggests that patient education is feasible and valuable in terms of improvements in quality of life, in function, in well-being and improved coping . Accordingly, guidelines recommend education and exercise as a core treatment for osteoarthritis.

Since 1994, Primary Health Care in Malmö has used a patient education programme directed towards OA.The program does not include exercise. In 2007-09 a study was made to investigate this education program.The study showed improvements in self-perceived health and in a few functional tests but not in self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis

Exclusion Criteria:

* Must be able to speak and understand swedish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Arthritis self-efficacy scale | at baseline
  Measure the patients self-efficacy
One-leg rising from sitting to standing | at baseline
  measure the strength
Grip Ability Test | at baseline
  Measure function of the hand
QuickDash | at baseline
  Measure self-percieved function of the arm/hand
Arthritis self-efficacy scale | after 4 month
  Measure the patients self-efficacy
One leg rising from sitting to standing | after 4 month
  measure the strength
Grip Ability Test | after 4 month
  Measure function of the hand
QuickDash | after 4 month
  Measure self-percieved function of the arm/hand

SECONDARY OUTCOMES:
Bipedal rising from sitting to standing | at baseline
  Measure the strength
One-legged jump | at baseline
  measure strength and balance
Standing on one leg with eyes open and standing on one leg with eyes closed | at baseline
  Measure the balance
Jamar | at baseline
  Measure the handstrength
PinchGauge | at baseline
  Measure the fingers strength
EQ5D | at baseline
  Measure self-percieved health
Bipedal rising from sitting to standing | after 4 month
  measure the strength
One-legged jump | after 4 month
  measure strength and balance
Standing on one leg with eyes open and standing on one leg with eyes closed | after 4 month
  measure the balance
Jamar | after 4 month
  Measure the handstrength
PinchGauge | after 4 month
  Measure the fingers strength
EQ5D | after 4 month
  Measure self-percieved health

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jönsson Lundgren, RPT, Principal Investigator — Lund University
Locations (1):
- Primary Health Care, Malmo, Skåne County, Sweden